CLINICAL TRIAL: NCT03314077
Title: Quality Control and Evaluation in Standard COPD Management
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Collaborators: Affiliated hospital of Guilin medical university,China (Unknown); University hospital of Hubei university for nationalities,China (Unknown); TongjiChibi hospital,China (Unknown); Central health center in Yongjiahe Town,China (Unknown); Chinses PLA general hospital (Unknown); Second Xiangya Hospital of Central South University (Other); the fourth affiliated hospital, Zhejiang university school of medcine (Unknown); First Hospital of China Medical University (Other); Peking University Third Hospital (Other); Huashan Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Shanghai Zhongshan Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); Yiwu Central Hospital (Other); Shanghai Xuhui Central Hospital (Unknown); Sijing hospital of Songjiang District in Shanghai (Unknown); Youxian People's Hospital (Unknown); Tong Ren hospital Shanghai Jiao Tong university school of medicine (Unknown); Zhejiang Putuo Hospital (Unknown); Jing-An District Center Hospital of Shanghai (Huashan Hospital Fudan University Jing-An Branch), Shanghai Medical College, Fudan University (Unknown)
Responsible Party: Principal Investigator, Weining Xiong, Professor, Tongji Hospital
Other Study IDs: TongjiHospitalResp.
Record Dates: First submitted 2017-10-15; First posted 2017-10-19 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard managed subjects: COPD patients accepted standard COPD management.
  Interventions: Other: GOLD 2017
- Controls: COPD patients didn't accepted standard COPD management or quality control, who are from hospital subjects with a retrospective cohort study.

INTERVENTIONS:
Other: GOLD 2017 — Standard COPD management according to GOLD 2017, and control the quality of management in one-year follow-up.
  Groups: Standard managed subjects

SUMMARY:
There is lack of quality control and evaluation indexes for standard COPD management in hospitals in China, leading to nonstandard in COPD management and discrepancy in therapeutic efficiency. This study focuses on establishing quality control and evaluation indexes for standard COPD management in hospitals in China, and evaluating the therapeutic efficiency after standard COPD management. This part is a prospective cohort which lasts 2 years. After standard COPD management according to GOLD 2017 by doctors in hospitals in China, patients will be followed up for their outcome after 1 year. Several indexes will be selected to evaluate the quality control of standard COPD management and its efficiency. The controls are from hospital-based subjects with a retrospective cohort study.

ELIGIBILITY:
Inclusion Criteria:

* 1.Clinical manifestation of COPD; post bronchodilator FEV1/FVC<0.70

Exclusion Criteria:

* 1. lung cancer. 2. Any history of psychiatric disorders. 3.HIV positive. 4.Breastfeeding, pregnancy or planning to be pregnant. 5.Estimated lifetime less than 1 years due to underlying diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinic-based population
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in spirometry | 1 years
  Spirometry will be assessed at baseline and through study completion

SECONDARY OUTCOMES:
Morbidity of acute exacerbation in 1 years | 1 year
  Morbidity of acute exacerbation completion will be assessed at baseline and through study

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - TongjiChibi hospital, Chibi, Hubei
  - Tongji hospital, Wuhan, Hubei